CLINICAL TRIAL: NCT05875233
Title: An Open-Label, 2-armed Study to Evaluate the Effect of Elix Cycle Balance and Daily Harmony on Polycystic Ovary Syndrome
Brief Title: A Study to Evaluate the Effect of Elix Cycle Balance and Daily Harmony on Polycystic Ovary Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zenchi, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 20318
Record Dates: First submitted 2023-04-19; First posted 2023-05-25 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Population will be split into 2 arms of 35 participants each: 1 group who are on hormonal birth control, and 1 group who are not on hormonal birth control. All participants will take the test product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group One: PCOS & Hormonal Birth Control (Active Comparator): All participants will have a diagnosis of PCOS and be regularly taking hormonal birth control.
  Interventions: Other: Elix Daily Harmony; Other: Elix Cycle Balance
- Group Two: PCOS with No Hormonal Birth Control (Active Comparator): All participants will have a diagnosis of PCOS and must not be taking any hormonal birth control.
  Interventions: Other: Elix Daily Harmony; Other: Elix Cycle Balance

INTERVENTIONS:
Other: Elix Daily Harmony — Elix Daily Harmony is a clinical-strength, organic blend of hormone-balancing Traditional Chinese Medicine (TCM) herbs and adaptogens. Contains Angelica Sinensis, licorice, ginger, Bupleurum, Cyperus Rotundus, White Peony, Mint, Poria, Atractylodes, White Ginseng, Reishi, Rehmannia Root, and Astragalus.
  Participants should add 3 droppers full (half a teaspoon or 2.5 ml) of Elix Daily Harmony to their tea or other warm or room temperature beverage each morning, 1-2 hours after their first meal. The product should not be taken with iced drinks or with food.
Other: Elix Cycle Balance — A tailored blend of medicinal herbs to holistically support menstrual symptoms by treating underlying imbalances. Participants should take 3 droppers full (half a teaspoon or 2.5 ml) of Elix Cycle Balance daily before bed with tea or other warm or room temperature beverage. The product should not be taken with iced drinks or with food.

SUMMARY:
This is a virtual, open-label, 2-armed study that will last 6 months. All participants will take the supplements daily and complete questionnaires at baseline and at the end of weeks 4, 8, 12, 16, 20, and 24 (study may be concluded at week 20 if results are seen earlier). The study will involve 70 participants with polycystic ovary syndrome (PCOS), 35 who are on hormonal birth control, and 35 who are not.

A subgroup of 20 participants from the non-birth control group, who experience hormonal acne/frequent hormonal breakouts will provide photographs of the face for expert skin grading at baseline, week 12, week 20, and week 24 (if the study is continued until week 24).

Questionnaires will be used to monitor changes in the menstrual cycle (regularity, frequency, predictability), bloating, fluid retention, weight gain, mood (mood swings, anxiety, mental clarity/focus, brain fog), pain, fatigue, acne, facial/bodily hair, and sleep quality. Expert skin grading will be carried out by a dermatologist to monitor changes in acne and skin clarity indicative of systemic effects of androgen excess. Likert scale responses will be statistically compared from baseline to each check-in. Participant responses on product feedback will be presented as % scores.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-36
* Diagnosed with PCOS in the last 5 years.
* Has experienced at least two of the following:

  1. Irregular menstrual periods or the absence of menstrual periods.
  2. Excessive facial or body hair, thinning hair, or hair loss on the scalp, oily skin, and or acne.
  3. Polycystic ovaries as determined by ultrasound.
* Otherwise generally healthy (not living with any uncontrolled chronic disease)
* Has concerns about irregular menstrual cycles and ovulation, mood swings, stress, tender breasts, food cravings, irritability, or low energy.
* Following stable, consistent diet and exercise regimens, and willing to refrain from making any lifestyle changes that may affect their menstrual cycle for the duration of the study.
* Willing to refrain from taking any other supplements that may target the menstrual cycle throughout the study period.
* Willing and able to adhere to the study protocol, including taking supplements at the required times, completing questionnaires via the technology portal, and where appropriate sharing the required photographs.
* Able to communicate in English.
* Participants must provide written informed consent (ICF).
* For the hormonal birth control group: must have been on the same hormonal birth control for the past 3 months and be willing to not make any changes to their hormonal birth control for the next 6 months.
* For the non-hormonal birth control group: must have been off hormonal birth control for the past 3 months and be willing to stay off hormonal birth control for the next 6 months.
* For the non-hormonal birth control group: Experience hormonal acne or frequent acne breakouts (a symptom of androgen excess).

Exclusion Criteria:

* Any pre-existing, unstable or uncontrolled medical or psychiatric illness.
* Anyone who has been diagnosed with endometriosis, uterine fibroids, pelvic inflammatory disease, reproductive cancers, chronic liver disease, diverticular disease, colorectal cancer or previous history of colorectal cancer, chronic pancreatitis, adenomyosis, fibromyalgia, rheumatoid arthiritis, lupus, inflammatory bowel disease, diagnosed chronic uncontrolled migraines, chronic pelvic pain syndrome, multiple sclerosis, chronic fatigue syndrome.
* Anyone who has undergone a hysterectomy, bilateral salpingo-oophorectomy, or any other gynecological medical or surgical treatment in the past 6 months.
* Anyone with significant abnormalities in the physical or laboratory examination. This includes having renal or liver function more than twice the normal range.
* Anyone with known severe allergic reactions that require the use of an epi-pen, or anyone who has any known allergy to any of the test product ingredients.
* Women who are pregnant, breastfeeding or attempting to become pregnant.
* Unwilling or unable to follow the study protocol.
* Users of any medication, herbal remedy, or supplement that can affect the menstrual cycle, or anyone who has used Elix Daily Harmony or Cycle Balance in the past.
* Anyone who has introduced a new medication, supplement or herbal remedies that target weight, skin (acne), mood, or menstrual cycle, in the last 3 months.
* Smokers, or anyone who has smoked in the past 6 months.
* Anyone with a history of substance abuse.
* Anyone who has more than 3 alcoholic drinks per day.
* Anyone with a BMI >35.
* For the hormonal birth control group: anyone who has changed their hormonal birth control in the past 3 months, or who is planning to change it in the next 6 months.
* For the non-hormonal birth control group: anyone who has been on hormonal birth control for the past 3 months, or who is planning to start using hormonal birth control in the next 6 months.

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-04-13 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of Daily Harmony and Elix Cycle Balance on menstrual cycle regularity and frequency. [Time Frame: Baseline to Week 24] | 24 weeks.
  Menstrual cycle frequency and regularity will be measured via self-reported questionnaire
To examine the effect of Daily Harmony and Elix Cycle Balance on acne as a symptom of hyperandrogenism. [Time Frame: Baseline to Week 24] | 24 weeks
  Assessed via self-reported questionnaires using the validated acne quality-of-life scale. Participants will record their score using a 7-point Likert Scale, with 1 representing the most severe symptoms and 7 representing the least severe symptoms.
To examine the effect of Daily Harmony and Elix Cycle Balance on acne measure via expert skin grading. [Time Frame: Baseline to Week 24] | 24 weeks
  Expert skin grading at baseline and at the end of weeks 12, 20, and 24 will be carried out by a dermatologist and used as a digital biomarker to evaluate improvements in PCOS related skin health (acne/skin clarity).

SECONDARY OUTCOMES:
To examine the effect of Daily Harmony and Elix Cycle Balance on PCOS-associated symptoms. [Time Frame: Baseline to Week 24] | 24 weeks
  Study-specific surveys will be used to assess the severity and incidence of common PCOS symptoms, including sleep quality bloating/fluid retention, weight gain, fatigue, mood swings, mental clarity/focus/brain fog, anxiety and pain. Participants will record their score using a 5-point Likert Scale, with 1 representing the most negative outcome and 5 representing the best outcome (no symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
TBC